CLINICAL TRIAL: NCT05423834
Title: Chronic Kidney Disease Progression in Chronic Hepatitis B Patients on Tenofovir Alafenamide (TAF) Versus Entecavir
Status: Active, not recruiting | Type: Observational
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lai Hung Wong, Professor, Chinese University of Hong Kong
Other Study IDs: TAF-renal study
Record Dates: First submitted 2022-06-13; First posted 2022-06-21 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Chronic Hepatitis B
MeSH Terms: conditions — Hepatitis B, Chronic | interventions — tenofovir alafenamide; entecavir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- TAF-treated Chronic hepatitis B patients: Chronic hepatitis B patients that treated with Tenofovir alafenamide
  Interventions: Drug: Tenofovir alafenamide
- ETV-treated Chronic hepatitis B patients: Chronic hepatitis B patients that treated with Entecavir
  Interventions: Drug: Entecavir

INTERVENTIONS:
Drug: Tenofovir alafenamide — Chronic hepatitis B patients who are receiving TAF as antiviral therapy for CHB, who were previously treatment naïve.
  Groups: TAF-treated Chronic hepatitis B patients
Drug: Entecavir — Chronic hepatitis B patients who are receiving ETV as antiviral therapy for CHB, who were previously treatment naïve.
  Groups: ETV-treated Chronic hepatitis B patients

SUMMARY:
Tenofovir alafenamide (TAF), a novel prodrug of tenofovir (TFV), has been approved for the treatment of chronic hepatitis B virus (HBV) infection. TAF has been shown to be a potent inhibitor of HBV replication at a low dose, with high intracellular concentration and more than 90% lower systemic TFV concentration than tenofovir disoproxil fumarate (TDF). TAF has been approved in the clinical practice guidelines in the west. Since its availability in Asia in 2017, there have been evolving data concerning its positive impact on renal safety as shown in registration trials.

The primary objective of this study is to compare the risk of chronic kidney disease (CKD) progression in chronic hepatitis B patients on TAF versus ETV in a territory-wide cohort in Hong Kong.

DETAILED DESCRIPTION:
Antiviral therapy with nucleos(t)ide analogues (NAs) has revolutionized the management of chronic hepatitis B (CHB) in the last two decades.1 Entecavir (ETV), a nucleoside analogue, is one of the first-line NAs recommended by all international treatment guidelines.2-4 As hepatitis B surface antigen (HBsAg) seroclearance rarely occurs, most patients require long-term, if not life-long, NA therapy. Hence, the safety of NAs requires careful scrutiny. In clinical trials, nephrotoxicity may occur in a small proportion of patients receiving nucleotide analogues. We previously demonstrated that tenofovir disoproxil fumarate (TDF) was associated with mild renal impairment in a minority of patients; those treated with entecavir (ETV) had a similar risk compared to untreated patients.5

Tenofovir alafenamide (TAF), a novel prodrug of tenofovir (TFV), has been approved for the treatment of chronic hepatitis B virus (HBV) infection. TAF has been shown to be a potent inhibitor of HBV replication at a low dose, with high intracellular concentration and more than 90% lower systemic TFV concentration than tenofovir disoproxil fumarate (TDF). TAF has been approved in the clinical practice guidelines in the west. Since its availability in Asia in 2017, there have been evolving data concerning its positive impact on renal safety as shown in registration trials.

ELIGIBILITY:
Inclusion Criteria:

* Positive hepatitis B surface antigen (HBsAg) or documented history of CHB for 6 months or more; AND
* On TAF 25 mg daily as antiviral treatment for CHB (cases); OR
* On ETV 0.5 to 1.0 mg daily as antiviral treatment for CHB (controls)

Exclusion Criteria:

* Previous NA treatment prior to TAF or ETV
* Positive antibody against hepatitis C, D, or human immunodeficiency virus (anti-HCV, anti-HDV, or anti-HIV)
* Evidence of other autoimmune or metabolic liver diseases (except non-alcoholic fatty liver disease).
* Moribund state including advanced/pre-terminal liver cancer or other non-hepatic cancers
* Non-hepatic cancer undergoing chemotherapy within last 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CHB patients who are receiving TAF or ETV as antiviral therapy for CHB, who were either previously treatment naïve.
Sampling Method: Probability Sample
Enrollment: 1800 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2025-12-21 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
CKD at 12 months | 12 months
  To evaluate chronic kidney disease (CKD) progression at 12 months. The CKD progression is defined as an increase in CKD stage for at least 1 stage for at least 3 consecutive months during follow-up.

SECONDARY OUTCOMES:
Change in eGFR | 12 months
  calculated using the CKD Epidemiology Collaboration (CKD-EPI) equation expressed as a single equation: GFR (in mL/min/1.73 m2) = 141 × min (Scr /κ, 1)α × max(Scr /κ, 1)-1.209 × 0.993Age × 1.018 [for the cases of females] × 1.159 [for the cases of ethnic Africans ]; where: Scr is the serum creatinine in mg/dL (equals to serum creatinine in micromole/L /88.4) , κ is 0.7 for females and 0.9 for males, α is -0.329 for females and -0.411 for males, min indicates the minimum of Scr /κ or 1, and max indicates the maximum of Scr /κ or 1.11 CKD stages 1, 2, 3A, 3B, 4 and 5 were defined based on eGFR

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Lo AO, Wong GL. Current developments in nucleoside/nucleotide analogues for hepatitis B. Expert Rev Gastroenterol Hepatol. 2014 Aug;8(6):607-22. doi: 10.1586/17474124.2014.909724. Epub 2014 Apr 30. PMID 24787673
- [Result] European Association for the Study of the Liver. EASL 2017 Clinical Practice Guidelines on the management of hepatitis B virus infection. J Hepatol. 2017 Aug;67(2):370-398. doi: 10.1016/j.jhep.2017.03.021. Epub 2017 Apr 18. PMID 28427875
- [Result] Sarin SK, Kumar M, Lau GK, Abbas Z, Chan HL, Chen CJ, Chen DS, Chen HL, Chen PJ, Chien RN, Dokmeci AK, Gane E, Hou JL, Jafri W, Jia J, Kim JH, Lai CL, Lee HC, Lim SG, Liu CJ, Locarnini S, Al Mahtab M, Mohamed R, Omata M, Park J, Piratvisuth T, Sharma BC, Sollano J, Wang FS, Wei L, Yuen MF, Zheng SS, Kao JH. Asian-Pacific clinical practice guidelines on the management of hepatitis B: a 2015 update. Hepatol Int. 2016 Jan;10(1):1-98. doi: 10.1007/s12072-015-9675-4. Epub 2015 Nov 13. PMID 26563120
- [Result] Terrault NA, Bzowej NH, Chang KM, Hwang JP, Jonas MM, Murad MH; American Association for the Study of Liver Diseases. AASLD guidelines for treatment of chronic hepatitis B. Hepatology. 2016 Jan;63(1):261-83. doi: 10.1002/hep.28156. Epub 2015 Nov 13. No abstract available. PMID 26566064
- [Result] Wong GL, Chan HL, Tse YK, Yip TC, Lam KL, Lui GC, Szeto CC, Wong VW. Chronic kidney disease progression in patients with chronic hepatitis B on tenofovir, entecavir, or no treatment. Aliment Pharmacol Ther. 2018 Nov;48(9):984-992. doi: 10.1111/apt.14945. Epub 2018 Aug 20. PMID 30125952